CLINICAL TRIAL: NCT04720625
Title: Adapt2Quit - A Machine-Learning, Adaptive Motivational System: RCT for Socio-Economically Disadvantaged Smokers
Brief Title: Adapt2Quit - An Adaptive Motivational System for Socio-Economically Disadvantaged Smokers
Acronym: A2Q
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Johns Hopkins University (Other); Baystate Health (Other)
Responsible Party: Principal Investigator, Rajani Sadasivam, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H00018991; 1R01CA240551-01A1 (NIH)
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After completing the screening, informed consent, and baseline data collection, study staff will enter the participant identification number and participant mobile phone number from the survey into an online system, and the system will assign allocation based on the randomization table. Using this technique, both smokers and the staff will be blinded to allocation during the initial session. Then, the research staff will be un-blinded to provide personalized training for intervention and control (note that staff who complete follow-up will be different and blinded to group assignment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapt2Quit (Experimental): These participants will receive Adapt2Quit motivational messaging and quitline facilitation messaging for 6 months.
  Interventions: Behavioral: Adapt2Quit
- Control (Active Comparator): These participants will receive quitline facilitation-only messaging for 6 months.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Adapt2Quit — Motivational text messages and quitline facilitation text messages will be sent to participants; these participants will receive Adapt2Quit (experimental) messages as well as quitline facilitation messages.
  Arms: Adapt2Quit
Behavioral: Control — Quitline facilitation text messages will be sent to participants; these participants will receive quitline facilitation-only messages.
  Arms: Control

SUMMARY:
The goal of this research is to test the Adapt2Quit computer program that uses participant input (message rating on how much the text motivational message might influence one to quit smoking) to select and text motivational messages that are more likely to help a user stop smoking. This Adapt2Quit system will be compared with a quitline facilitation-only control (text messages will be sent to facilitate quitline use). The primary research hypothesis is that the Adapt2Quit recommender-selected messages will be more effective than a texting quitline facilitation-only control for smoking cessation among socioeconomically disadvantaged (SED) smokers.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker
* Socioeconomically disadvantaged (SED) (using the following criteria: unemployed or underemployed, low income as defined by the federal poverty level guidelines, uninsured or underinsured, and/or have less than a high school education)
* English-speaking
* Active in care (at least two clinical visits in the last year)
* Have a texting-enabled cell phone

Exclusion Criteria:

* Not a current smoker
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Pregnant women
* Pilot study participants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Self-Reported Participant Tobacco Cessation Rate (quit rate) | 6-months post-randomization
  Self-reported 6-month point prevalence cessation (yes/no) will be assessed at 6-month follow-up.
Biochemical Carbon Monoxide (CO) Verification of Tobacco Cessation | 6-months post-randomization
  Biochemical carbon monoxide (CO) verification testing will also be done for a small subset of participants, where 0-6 parts per million (PPM) measures a non-smoker and 7+ PPM indicates a current smoker.

SECONDARY OUTCOMES:
Time to First Quit Attempt | From randomization to 6-months post-randomization
  Self-reported date of first quit attempt since starting the study will be assessed through text message response from participant during the 6-month intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Rajani Sadasivam, PhD, Principal Investigator — Associate Professor
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamberi A, Weitz B, Flahive J, Eve J, Najjar R, Liaghat T, Ford D, Lindenauer P, Person S, Houston TK, Gauvey-Kern ME, Lobien J, Sadasivam RS, Balakrishnan K. Testing a Machine Learning-Based Adaptive Motivational System for Socioeconomically Disadvantaged Smokers (Adapt2Quit): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 16;14:e63693. doi: 10.2196/63693. PMID 40239194